CLINICAL TRIAL: NCT07264062
Title: Optimizing Care to Prevent Diabetes and Promote Cardiovascular Health Among Younger Adults With Severe Mental Illness
Brief Title: MetSense Pilot and Feasibility
Acronym: MetSenseP&F
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Esti Iturralde, Research Scientist I, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1850120-11; K23MH126078 (NIH)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Serious Mental Illness; Type 2 Diabetes
Keywords: serious mental illness; type 2 diabetes; diabetes prevention; prediction model; clinical decision support
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 2-arm pragmatic cluster-randomized pilot feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MetSense (Active Comparator): Participants will be managed by clinical pharmacists who are able to view the MetSense risk flag.
  Interventions: Behavioral: MetSense Risk Flag
- Usual Care (Other): Participants will receive usual care. They will be managed by clinical pharmacists who are not able to view the MetSense risk flag.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: MetSense Risk Flag — The MetSense risk flag alerts the clinician if the patient has high diabetes risk and prompts additional diabetes risk management.
  Arms: MetSense
Other: Usual Care — Participants will receive usual care.
  Arms: Usual Care

SUMMARY:
People with serious mental illness have high risk for type 2 diabetes due to multiple risk factors, including the metabolic side effects of psychotropic medications that are used to treat these conditions. Type 2 diabetes is preventable through lifestyle and pharmacological interventions, but many people with serious mental illness do not receive regular screening for type 2 diabetes risk. In many health care settings, clinical pharmacists are increasingly managing patients with serious mental illness and have expertise in monitoring the metabolic side effects of psychotropic medications. This study evaluates the feasibility and acceptability of using a diabetes prediction model that is based on electronic health record data (the MetSense risk flag) to alert clinical pharmacists about patients who are at high diabetes risk, prompting these clinicians to prioritize diabetes risk management services.

DETAILED DESCRIPTION:
MetSense is a clinical decision support tool that is being developed to help clinicians prioritize diabetes risk management services for patients with serious mental illness who have high diabetes risk. This study seeks to evaluate the feasibility, acceptability, and preliminary effectiveness of using the MetSense risk flag to prompt further evaluation of metabolic risk factors and to prioritize other diabetes risk management services, including diabetes risk screening, care coordination with patients' primary care physicians, and pharmacological management of diabetes risk. In this pragmatic, cluster-randomized trial, patients with serious mental illness will be allocated to 1 of 2 trial arms based on which clinical pharmacist manages their care. The clinical pharmacists will be randomized to view the MetSense risk flag (intervention arm) or to not view the MetSense risk flag (control arm, i.e., usual care). The primary outcome is completion of hemoglobin A1c laboratory testing. The study will also examine differences in clinician evaluation of metabolic risk factors, body mass index measurement, prediabetes diagnosis, diabetes diagnosis, primary care visits, metformin medication dispensing, hemoglobin A1c result, body mass index result, and clinician-reported acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with schizophrenia, another psychotic disorder, or bipolar disorder
* Included in a clinical pharmacist population management program for serious mental illness within Kaiser Permanente Northern California

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent with completed hemoglobin A1c test within 6 months. | 6 months
  Laboratory test completion

SECONDARY OUTCOMES:
Percent with clinician evaluation of metabolic risk factors as documented in the electronic health record within 6 months. | 6 months
  Electronic health record documentation via smartphrase
Percent with body mass index measurement within 6 months. | 6 months
  Body mass index recorded in the electronic health record
Percent with prediabetes diagnosis within 6 months. | 6 months
  Diagnosis documented in the electronic health record
Percent who attended a primary care visit within 6 months. | 6 months
  Visit documented in the electronic health record
Percent with metformin medication dispensed within 6 months. | 6 months
  Dispensing based on pharmacy records
Average hemoglobin A1c value based on the final measurement in 6 months. | 6 months
  Laboratory value
Average body mass index based on the final measurement in 6 months. | 6 months
  Value recorded in the electronic health record

OTHER OUTCOMES:
Average clinician acceptability score at 6 weeks. | 6 weeks
  Questionnaires and qualitative interview
Average clinician acceptability score at 10 weeks. | 10 weeks
  Questionnaires and qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Esti Iturralde, PhD, Principal Investigator — KPNC Division of Research
Locations (1):
- KPNC Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iturralde E, Fazzolari L, Shia M, Slama N, Leang J, Awsare S, Nguyen LT. Closing the Care Gap for People with Severe and Persistent Mental Illness: Collaborative Care, Telehealth, and Clinical Pharmacy. NEJM Catal Innov Care Deliv. 2022 May;3(5):10.1056/CAT.21.0417. doi: 10.1056/CAT.21.0417. PMID 36569369
- [Background] Iturralde E, Fazzolari L, Slama NE, Alexeeff SE, Sterling SA, Awsare S, Koshy MT, Shia M. Telehealth Collaborative Care Led by Clinical Pharmacists for People With Psychosis or Bipolar Disorder: A Propensity Weighted Comparison With Usual Psychiatric Care. J Clin Psychiatry. 2024 Jan 29;85(1):23m14917. doi: 10.4088/JCP.23m14917. PMID 38301189